CLINICAL TRIAL: NCT00002047
Title: Retrovir Capsules in the Treatment of HIV-Infected Patients in Renal Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 014H; 27433-19
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1990-05

CONDITIONS: HIV Infections; Kidney Failure, Chronic
Keywords: Kidney Failure, Chronic; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Zidovudine; Renal Dialysis
MeSH Terms: conditions — HIV Infections; Kidney Failure, Chronic; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Zidovudine

INTERVENTIONS:
Drug: Zidovudine

SUMMARY:
To evaluate the safety, tolerance, and pharmacokinetics of Retrovir (AZT) administration in HIV-infected patients in renal failure receiving maintenance hemodialysis.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* A positive HIV antibody test (ELISA confirmed by Western blot).
* Chronic renal failure managed by a stable hemodialysis regimen.
* Acceptable hepatic function defined by specified lab values.
* Life expectancy > 6 months.
* Enrollment is limited to 9 chronic hemodialysis patients and 9 Continuous Ambulatory Peritoneal Dialysis (CAPD) patients. These patients must be stable in their ESRD treatment regimen before entry.

Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* Active, serious opportunistic infections at the time of study entry.
* Fever > 100 degrees F at study entry.
* Severe malabsorption (evidenced by persistent diarrhea of greater than 4 weeks duration with = or > 6 loose stools per day accompanied by significant weight loss).

Patients with the following are excluded:

* Active, serious opportunistic infections at the time of study entry.
* Fever > 100 degrees F at study entry.
* Severe malabsorption (evidenced by persistent diarrhea of greater than 4 weeks duration with = or > 6 loose stools per day accompanied by significant weight loss).

Prior Medication:

Excluded within 2 weeks of study entry:

- Any other experimental therapy. Drugs which cause significant bone marrow suppression. Rifampin or rifampin derivatives. Cytolytic chemotherapy. Drugs which cause significant hepatotoxicity.

Excluded within 4 weeks of study entry:

- Immunomodulating agents, including steroids, interferon, Isoprinosine, and interleukin 2.

Excluded within 8 weeks of study entry:

- Other antiretroviral agents (e.g., zidovudine [AZT], suramin, ribavirin, HPA-23, foscarnet, dextran sulfate, disulfiram, ddA/ddC, or dideoxycytidine).

Active drug or alcohol abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Univ of Maryland at Baltimore, Baltimore, Maryland, United States